CLINICAL TRIAL: NCT04196439
Title: Comparison Of Continuous Epidural Analgesia And Ultrasound Guided Continuous Supra-Inguinal Fascia Iliaca Compartment Block After Total Hip Replacement Surgery
Brief Title: Continuous Epidural Analgesia Versus Continuous Supra-Inguinal Fascia Iliaca Block in Total Hip Replacement Surgery
Acronym: S-FICB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmad Samir Alabd, assistant lecturer of anaesthesiology, Master degree, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: supra-inguinal fascia iliaca
Record Dates: First submitted 2019-11-01; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- continuous epidural analgesia (Active Comparator): continuous lumbar epidural catheter inserted preoperatively before induction of general anaesthesia
  Interventions: Procedure: continuous epidural analgesia
- continuous supra-inguinal fascia iliaca compartment block (Active Comparator): ultrasound guided supra-inguinal FICB with insertion of catheter for continuous infusion before induction of general anaesthesia.
  Interventions: Procedure: supra-inguinal fascia iliaca compartment block

INTERVENTIONS:
Procedure: continuous epidural analgesia — injection of local anaesthetic into epidural space
  Other Names: continuous epidural anaesthesia
  Arms: continuous epidural analgesia
Procedure: supra-inguinal fascia iliaca compartment block — ultrasound guided injection of local anaesthetic into fascia iliaca compartment
  Other Names: Supra-inguinal FICB
  Arms: continuous supra-inguinal fascia iliaca compartment block

SUMMARY:
comparison of continuous epidural analgesia and ultrasound guided continuous supra-inguinal fascia iliaca compartment block after total hip replacement surgery

DETAILED DESCRIPTION:
supra-inguinal FICB is a promising safe approach for lumbar plexus that may be useful for analgesia in hip surgeries.In this study the investigators are comparing continuous S-FICB with continuous epidural analgesia after total hip arthroplasty surgeries with the primary aim to assess efficacy of post-operative analgesia, and secondary aim to assess rehabilitation indices, side effects and radiological pattern of local anaesthetic distribution after S-FICB.

ELIGIBILITY:
Inclusion Criteria:

* orthopaedic patients, American Society of Anesthesiologists (ASA) physical status I-III, scheduled to undergo unilateral total hip replacement surgery via lateral approach

Exclusion Criteria:

* 1- History of neurological/neuromuscular, psychiatric disease, dementia preventing proper comprehension.

  2- Patients younger than 18 years or older than 80 years. 3- Patients with Body Mass Index (BMI) <18.5 or >30 kg/m2. 4- Coagulation disturbances (INR>1.4, platelet count<100 000). 5- History of opioid dependence (opioid use within the last 4 weeks). 6- History of allergies to study medications. 7- Other contraindications to neuraxial blockade (e.g., patient refusal, local/systemic sepsis, low fixed cardiac output).

  8- Contraindications to continuous fascia iliaca compartment block (e.g., infection overlying the injection site or previous femoro-popliteal bypass surgery).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-02 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
postoperative analgesia after THA surgery | 36 hours
  visual analogue scale (VAS) scores for pain assessment at rest and movements and morphine consumption

SECONDARY OUTCOMES:
radiological pattern of local anaesthetic distribution in S-FICB group | 30 minutes after local anaesthetic injection
  imaging of pelvis using x-rays c arm machine
success of rehabilitation | 36 hours
  rehabilitation indices achievement after THA

CONTACTS AND LOCATIONS:
Overall Officials: Emad A Abdelmonem, M.D., Study Chair — Alexandria faculty of medicine
Locations (1):
- Alexandria faculty of medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vermeylen K, Desmet M, Leunen I, Soetens F, Neyrinck A, Carens D, Caerts B, Seynaeve P, Hadzic A, Van de Velde M. Supra-inguinal injection for fascia iliaca compartment block results in more consistent spread towards the lumbar plexus than an infra-inguinal injection: a volunteer study. Reg Anesth Pain Med. 2019 Feb 22:rapm-2018-100092. doi: 10.1136/rapm-2018-100092. Online ahead of print. PMID 30798268
- [Background] Hebbard P, Ivanusic J, Sha S. Ultrasound-guided supra-inguinal fascia iliaca block: a cadaveric evaluation of a novel approach. Anaesthesia. 2011 Apr;66(4):300-5. doi: 10.1111/j.1365-2044.2011.06628.x. Epub 2011 Feb 24. PMID 21401544
- [Background] Vermeylen K, Soetens F, Leunen I, Hadzic A, Van Boxtael S, Pomes J, Prats-Galino A, Van de Velde M, Neyrinck A, Sala-Blanch X. The effect of the volume of supra-inguinal injected solution on the spread of the injectate under the fascia iliaca: a preliminary study. J Anesth. 2018 Dec;32(6):908-913. doi: 10.1007/s00540-018-2558-9. Epub 2018 Sep 24. PMID 30250982
- [Background] Bullock WM, Yalamuri SM, Gregory SH, Auyong DB, Grant SA. Ultrasound-Guided Suprainguinal Fascia Iliaca Technique Provides Benefit as an Analgesic Adjunct for Patients Undergoing Total Hip Arthroplasty. J Ultrasound Med. 2017 Feb;36(2):433-438. doi: 10.7863/ultra.16.03012. Epub 2016 Dec 10. PMID 27943417
- [Background] Bang S, Chung J, Jeong J, Bak H, Kim D. Efficacy of ultrasound-guided fascia iliaca compartment block after hip hemiarthroplasty: A prospective, randomized trial. Medicine (Baltimore). 2016 Sep;95(39):e5018. doi: 10.1097/MD.0000000000005018. PMID 27684871